CLINICAL TRIAL: NCT06265363
Title: Evaluation of the Frequency of Retinopathy of Prematurity, Influencing Risk Factors, and Treatment Outcomes in Premature Infants with a Birth Weight >1500 Grams or Gestational Age ≥33 Weeks in Turkey.
Brief Title: Evaluation of the Frequency, Risk Factors, and Outcomes of ROP in Infants with a BW >1500 Grs or GA ≥33 Wks in Turkey.
Acronym: TR-ROP-2
Status: Recruiting | Type: Observational
Sponsor: Baskent University Ankara Hospital (Other)
Collaborators: Hacettepe University (Other); Gazi University (Other); Gaziosmanpasa Research and Education Hospital (Other Government); Celal Bayar University (Other); Selcuk University (Other); Recep Tayyip Erdogan University (Other); Karadeniz Technical University (Other); Istinye University (Other); Biruni University (Other); Ordu University (Other); Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government); Pamukkale University (Other); Kanuni Sultan Suleyman Training and Research Hospital (Other); Konya City Hospital (Other); Kecioren Education and Training Hospital (Other); Ataturk University (Other); Meda Hospital (Unknown); Eskisehir Osmangazi University (Other); Necmettin Erbakan University (Other); Kırıkkale University (Other); Sisli Hamidiye Etfal Training and Research Hospital (Other); Acibadem Atakent University Hospital (Other); Balikesir Ataturk City Hospital (Other Government); Kocaeli University (Other); Acibadem Maslak Hospital (Other); Erzurum City Hospital (Other); Afyon Karahisar Hospital (Unknown); Ankara Koru Hospital (Unknown); Gulhane School of Medicine (Other); Bursa Yuksek Ihtisas Training and Research Hospital (Other Government); Namik Kemal University (Other); Bursa City Hospital (Other Government); Kayseri City Hospital (Other Government); Ankara Etlik City Hospital (Other Government); Zonguldak Bulent Ecevit University (Other); Gazi Yasargil Training and Research Hospital (Unknown); Inonu University (Other); Dr. Behcet Uz Children's Hospital (Other); Ankara Training and Research Hospital (Other); Tepecik Training and Research Hospital (Other); Aydin Adnan Menderes University (Other); Dicle University (Other); Akdeniz University (Other); Umraniye Education and Research Hospital (Other Government); Ankara City Hospital Bilkent (Other); Afyonkarahisar University of Health Sciences Health Application and Research Center (Unknown); Harran University (Other); Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other); Istanbul University - Cerrahpasa (Other); Uludag University (Other); Sanliurfa Education and Research Hospital (Other Government); Dokuz Eylul University (Other); Bursa Doruk Yıldırım Hospital (Unknown); Malatya Turgut Ozal University (Other); Abant Izzet Baysal University (Other); Alanya Training and Research Hospital (Unknown); İstanbul Training and Research Hospital (Unknown); Baskent University (Other); Kahramanmaras Sutcu Imam University (Other); Batman Training and Research Hospital (Other Government); Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other); Acıbadem Atunizade Hospital (Other); Adiyaman Training and Research Hospital (Unknown); Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other); Ondokuz Mayıs University (Other); Trakya University (Other); Trabzon Kanuni Education and Research Hospital (Other); Seyhan Hospital (Unknown); Esenyurt University Hospital (Unknown); Başakşehir Çam & Sakura City Hospital (Other Government); Sakarya University (Other); Mardin Training and Research Hospital (Unknown); Karabuk University (Other); Giresun Training and Research Hospital (Unknown); Koc University Hospital (Other); Tekirdağ City Hospital (Unknown); Istanbul Medipol University Hospital (Other); Adana City Training and Research Hospital (Other); Istanbul University (Other); Marmara University Pendik Training and Research Hospital (Other); Medikal Park Ankara Hospital (Unknown); Muğla Sıtkı Koçman University (Other); Yuzuncu Yil University (Other); Sanko University (Other); Antalya Training and Research Hospital (Other Government); Firat University (Other); Ankara Guven Hospital (Unknown); Private Batman Hospital (Unknown); İstanbul Bağcılar Training and Research Hospital (Unknown); Istanbul Aydın University (Other); Mersin City Hospital (Unknown)
Responsible Party: Principal Investigator, Sezin Unal, Sezin Unal, MD, Baskent University Ankara Hospital
Other Study IDs: TR-ROP-2 Study
Record Dates: First submitted 2024-02-01; First posted 2024-02-20 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study includes preterm infants who are being screened for ROP between August 1,2023 and August 1, 2024 in 94 neonatal intensive care units (NICUs) in Turkey. Infants with birth weight (BW) of >1500 g or ≥ 33 weeks' gestation who are screened for retinopathy of prematurity are included. The incidence of any ROP, severe ROP and treatment modalities will be determined. The risk factors for ROP development will also be evaluated.

DETAILED DESCRIPTION:
This study, promoted by the "Turkish Neonatology Society", involved preterm infants who are being screened for ROP between August 1,2023 and August 1, 2024 in level III/IV Turkish NICUs.

An electronic questionnaire is being filled by certified neonatologists in Turkey via a special network. Neonatologists working in 94 centers who agreed to participate in this study provide their data regarding the ROP in their NICU. The medical records of retinal examinations of preterm infants who met the screening criteria will be evaluated.

A case report form for each patient will be filled including risk factors for the development of ROP such as gestational age, birth weight, small for gestational age (SGA), gender, multiple gestation, antenatal steroid therapy, invitro fertilization, preeclampsia/eclampsia, infants of diabetic mother, chorioamnionitis, resuscitation in delivery room, respiratory distress syndrome (RDS), duration of mechanical ventilation and oxygen therapy, intracranial hemorrhage, hemodynamically significant patent ductus arteriosus (PDA), early/late sepsis, necrotising enterocolitis (NEC), number of blood transfusions, bronchopulmonary dysplasia (BPD), time to full enteral feeding, percentage of own mothers milk.

Risk factors for developing ROP will be evaluated. Multivariate analysis will be performed among significant variables. In addition, the incidence of any ROP, severe ROP in relation to GA and BW and treatment modalities will be determined.

Severe ROP is defined as ROP requiring treatment. Since Turkey is receiving many refugees in recent years, the investigators also planned to evaluate the incidence and risk factors for developing ROP in preterm babies of refugees.

Ophthalmologic examination is continued until full vascularisation. So, the maximum stage of ROP detected for every infant will be reported. Data from 94 NICUs will be pooled together and analyzed.

The "International Classification of ROP" guidelines (ICROP-3) are used to record the stage of disease, location by zone, signs of plus disease and signs of regression/reactivation/persistent avascular retina.

Criteria for treatment of ROP are based on the Early Treatment for Retinopathy of Prematurity (ETROP) recommendation.

Confirmed forms are also assigned by the parents before the initial screening and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Infants with BW >1500 g or ≥33 weeks' gestation who were determined to be at risk for ROP by the attending clinician and were screened for ROP.

Exclusion Criteria:

* Neonates who died before the first ROP examination are excluded from the study.

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants with BW >1500 g or ≥33 weeks' gestation who were screened for ROP.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of ROP | 12 months
  Incidence of ROP and severe ROP in infants > 1500 gr and gestational age ≥ 33 weeks in Turkey.

SECONDARY OUTCOMES:
The role of being SGA in infants in the development of ROP | 12 months
  Number of infants with less than 10th percentile of birth weight according to Fenton graphs
The role of sepsis in infants in the development of ROP | 12 months
  Number of infants diagnosed with early sepsis (< 3 days postnatal) or late sepsis (>3 days postnatal) during the NICU admission
The role of mechanical ventilation in infants in the development of ROP | 12 months
  Duration of invasive mechanical ventilation during NICU admission
The role of chorioamnionitis in infants in the development of ROP | 12 months
  The number of infants whose mothers with clinical/histological chorioamnionitis
Laser photocoagulation treatment | 12 months
  Number of patients requiring laser photocoagulation treatment
Anti-VEGF treatment | 12 months
  Number of patients requiring anti-VEGF treatment
Vitreoretinal surgery | 12 months
  Number of patients requiring vitreoretinal surgery

CONTACTS AND LOCATIONS:
Overall Officials: Esin Koç, MD, Study Director — Gazi University; Ahmet Y Bas, MD, Study Director — Ankara Yildirim Beyazıt University; İbrahim M Hirfanoğlu, MD, PhD, Study Director — Gazi University; Sezin Unal, MD, Study Director — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiang MF, Quinn GE, Fielder AR, Ostmo SR, Paul Chan RV, Berrocal A, Binenbaum G, Blair M, Peter Campbell J, Capone A Jr, Chen Y, Dai S, Ells A, Fleck BW, Good WV, Elizabeth Hartnett M, Holmstrom G, Kusaka S, Kychenthal A, Lepore D, Lorenz B, Martinez-Castellanos MA, Ozdek S, Ademola-Popoola D, Reynolds JD, Shah PK, Shapiro M, Stahl A, Toth C, Vinekar A, Visser L, Wallace DK, Wu WC, Zhao P, Zin A. International Classification of Retinopathy of Prematurity, Third Edition. Ophthalmology. 2021 Oct;128(10):e51-e68. doi: 10.1016/j.ophtha.2021.05.031. Epub 2021 Jul 8. PMID 34247850
- [Background] Bas AY, Demirel N, Koc E, Ulubas Isik D, Hirfanoglu IM, Tunc T; TR-ROP Study Group. Incidence, risk factors and severity of retinopathy of prematurity in Turkey (TR-ROP study): a prospective, multicentre study in 69 neonatal intensive care units. Br J Ophthalmol. 2018 Dec;102(12):1711-1716. doi: 10.1136/bjophthalmol-2017-311789. Epub 2018 Mar 8. PMID 29519879
- [Background] Bas AY, Koc E, Dilmen U; ROP Neonatal Study Group. Incidence and severity of retinopathy of prematurity in Turkey. Br J Ophthalmol. 2015 Oct;99(10):1311-4. doi: 10.1136/bjophthalmol-2014-306286. Epub 2015 Apr 13. PMID 25868788